CLINICAL TRIAL: NCT01875705
Title: An Open-Label, Phase I, Dose-Escalation Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0994 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Dose-Escalation Study of GDC-0994 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GO28885; 2013-000566-10 (EudraCT Number)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — ravoxertinib

ARMS (2):
- Stage I-Dose Escalation (Experimental)
  Interventions: Drug: GDC-0994
- Stage II-Cohort-Expansion (Experimental)
  Interventions: Drug: GDC-0994

INTERVENTIONS:
Drug: GDC-0994 — Escalating doses of GDC-0994 until maximum tolerated dose is reached
  Arms: Stage I-Dose Escalation
Drug: GDC-0994 — Recommended dose determined in Stage I-Dose Escalation phase, until disease progression
  Arms: Stage II-Cohort-Expansion

SUMMARY:
This is an open-label, multicenter, dose-escalation study to assess the safety, tolerability, and pharmacokinetics of GDC-0994 in patients with locally advanced or metastatic solid tumors. Patients will be enrolled in one of two stages: a dose-escalation stage (Stage I) or the subsequent expansion stage (Stage II). Stage I will evaluate the safety, tolerability, and pharmacokinetics of increasing doses of GDC-0994 administered daily. Stage II will gather additional data on safety, tolerability, and pharmacokinetics of the recommended dose of GDC-0994 determined in Stage I.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically documented, locally advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable
* Evaluable disease or disease measurable per RECIST 1.1
* Life expectancy >= 12 weeks
* Adequate hematologic and end organ function
* Consent to provide archival tissue

Exclusion Criteria:

* History of prior significant toxicity from another MEK or ERK inhibitor requiring discontinuation of treatment
* History of parathyroid disorder or history or malignancy-associated hypercalcemia requiring therapy in the past 6 months
* Evidence of visible retinal pathology as assessed by ophthalmologic examination that is considered a risk factor for retinal vein thrombosis or neurosensory retinal detachment
* History of glaucoma
* Intraocular pressure > 21 mmHg as measured by tonometry
* Predisposing factors to retinal vein occlusion, including uncontrolled hypertension, uncontrolled diabetes, uncontrolled hyperlipidemia, and coagulopathy
* History of retinal vein occlusion (RVO), neurosensory retinal detachment, or neovascular macular degeneration
* Allergy or hypersensitivity to components of the GDC-0994 formulation
* Palliative radiotherapy within 2 weeks prior to first dose of study drug treatment in Cycle 1
* Experimental therapy within 4 weeks prior to first dose of study drug treatment in Cycle 1
* Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose of study drug treatment in Cycle 1, or anticipation of the need for major surgery during the course of study treatment
* Prior anti-cancer therapy within 28 days or 5 times the half-life whichever is longer
* Current severe, uncontrolled systemic disease
* History of clinically significant cardiac dysfunction
* Pregnancy, lactation, or breastfeeding
* Active autoimmune disease
* Inability or unwillingness to swallow pills
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* Clinically significant history of liver disease (including cirrhosis), current alcohol abuse, or current known active infection with HIV, hepatitis B virus, or hepatitis C virus
* Any condition requiring warfarin or thrombolytic anticoagulants
* Uncontrolled ascites requiring weekly large volume paracentesis for 3 consecutive weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | Approximately 2 years
Maximum tolerated dose | Approximately 2 years
Dose-limiting toxicities | Approximately 2 years
Pharmacokinetics: Area under the concentration-time curve | Approximately 2 years
Pharmacokinetics: Maximum plasma concentrations | Approximately 2 years
Pharmacokinetics: Minimum plasma concentrations | Approximately 2 years
Pharmacokinetics: Time to maximum plasma concentration | Approximately 2 years
Pharmacokinetics: Apparent terminal elimination half-life | Approximately 2 years

SECONDARY OUTCOMES:
To assess the PD effects of GDC-0994, as measured by changes in molecular biomarkers in pre- and post-treatment tumor tissues\n | Approximately 2 years
Objective Response according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Approximately 2 years
Progression-free survival according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Approximately 2 years
Duration of response according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (3):
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Karmanos Can Inst, Detroit, Michigan
  - Sarah Cannon Research Inst., Nashville, Tennessee
- Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif, France